CLINICAL TRIAL: NCT06394505
Title: Operating Room Nurses' Risks and Perceptions of Safety Climate
Status: Completed | Type: Observational
Sponsor: İslam Elagöz (Other)
Responsible Party: Sponsor-Investigator, İslam Elagöz, Director, Kilis 7 Aralik University
Organization: Kilis 7 Aralik University (Other)
Other Study IDs: kilis?_8
Record Dates: First submitted 2024-04-27; First posted 2024-05-01 (Actual); Last update posted 2024-05-02 (Actual); Status verified 2024-04

CONDITIONS: Safety Issues; Nursing Caries
Keywords: climate safety; nursing; operating room

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Data Collection Tools — Safety Climate Scale: Since a customized safety climate perception measurement tool for nurses could not be found in the literature, the "Safety Climate Scale" (SAS), developed by Choudry et al. in 2009 and adapted to Turkish by Türen et al. in 2014, was used on healthcare workers and electronics industry workers. The scale consists of two subscales: 10 items evaluating the management's perspective and rules (YÖBAK) and 4 items evaluating colleagues and safety training (İAGE). Participants rate the statements in the scale between "strongly agree" (five points) and "strongly disagree" (one point). The total score of the scale is calculated by taking the average of the item scores, and as the average gets closer to five, the safety climate improves, and as it gets closer to one, it gets worse. The Cronbach Alpha reliability coefficient of the scale was determined as 0.93 in the study conducted by Türen et al., and in this study it was calculated as 0.82.
  Other Names: Socio-Demographic Characteristics Survey Form:

SUMMARY:
One of the leading elements in providing safe healthcare is to maintain employee health and safety. Hazards in the working environments of healthcare professionals threaten employee safety and cause errors in patient care. In this case, healthcare professionals working in a safe environment means that patients receive service in a safe environment.

Safety climate is the perception of employees of the policies, procedures and practices that exist to ensure safety in the workplace and is an important element for the formation of a safety culture in the workplace. There are many factors that determine the perception of safety climate. These factors can be listed as the type and size of the organization, the occupational risks that employees are exposed to at work, the way occupational safety is managed, the gender, seniority of employees, and their position in the organization.

DETAILED DESCRIPTION:
An organization's safety culture and team members' perceptions of the safety climate influence patient safety outcomes. Measuring the safety climate in healthcare workplaces is important to monitor the change of safety culture in the workplace over time. In units with a high safety climate, the patient safety climate is also hi.

The extent to which employees believe in and embrace safety practices, policies and procedures is a reflection of the overall safety culture. A healthy climate plays an important role in increasing both the safety of employees and the safety of patients. According to AORN, the safety of the work environment equals patient safety. There are studies showing that the risks affecting operating room staff threaten patient safety . Therefore, it is necessary to analyze the safety environment in the operating room to improve patient safety.

Evaluating the opinions and perceptions of operating room staff is important in identifying and managing risks in the operating room and creating a safety culture. Because intense dynamics, constantly changing situations and high stress levels can make it difficult to create and maintain a positive safety climate in operating rooms. Therefore, operating room managers and healthcare organizations need to pay attention to employees' risk perceptions and safety climate assessments. Although WHO emphasizes the importance of ensuring safety and safety culture in operating rooms, problems continue to occur in this regard.

The purpose of this study is to determine the risks that operating room nurses encounter during their professional activities and to evaluate how these risks affect nurses' perceptions of safety climate.

ELIGIBILITY:
Inclusion Criteria:

* Having been working as an operating room nurse for at least one year in the hospitals where the research was conducted, Having actively worked in operating room duties during the research, Voluntarily expressing participation in the study.

Exclusion Criteria:

* Data from participants who took long-term leave during the study period or worked in a department other than the operating room, refused to start the study, or wanted to withdraw after starting the study were not taken into account in the final analysis

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Application of Research The research was conducted using an online survey. Operating room nurses were invited to the survey link via e-mail, and participation in the survey was voluntary. The survey includes socio-demographic information and the Security Climate Scale. The survey took approximately 15-20 minutes to complete.
Sampling Method: Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2024-03-01 (Actual); Primary Completion 2024-04-01 (Actual); Study Completion 2024-04-26 (Actual)

PRIMARY OUTCOMES:
Safety Climate Scale: | up to 4 weeks
  Since a customized safety climate perception measurement tool for nurses could not be found in the literature, the "Safety Climate Scale" (SAS), developed by Choudry et al. in 2009 and adapted to Turkish by Türen et al. in 2014, was used on healthcare workers and electronics industry workers. The scale consists of two subscales: 10 items evaluating the management's perspective and rules (YÖBAK) and 4 items evaluating colleagues and safety training (İAGE). Participants rate the statements in the scale between "strongly agree" (five points) and "strongly disagree" (one point). The total score of the scale is calculated by taking the average of the item scores, and as the average gets closer to five, the safety climate improves, and as it gets closer to one, it gets worse. The Cronbach Alpha reliability coefficient of the scale was determined as 0.93 in the study conducted by Türen et al., and in this study it was calculated as 0.82.

CONTACTS AND LOCATIONS:
Overall Officials: Kübra KAYA, PhD, Study Chair — devlet hastanesi
Locations (1):
- Islam, Kilis, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No